CLINICAL TRIAL: NCT04773457
Title: Neutrophil Phenotypic Profiling and Surgical Site Infections in Surgical Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00037804
Record Dates: First submitted 2021-02-12; First posted 2021-02-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-01

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spine Surgery: Pediatric patients presenting for elective spine fusion surgery at Boston Children's Hospital
  Interventions: Other: Surgical Site Infection
- Abdominal Surgery: Pediatric patients presenting for elective abdominal surgery at Boston Children's Hospital
  Interventions: Other: Surgical Site Infection

INTERVENTIONS:
Other: Surgical Site Infection — infection at the site of the surgery (spine or abdomen)

SUMMARY:
Surgical site infections (SSIs) are one of the major hospital acquired infections and responsible for the most cost among the hospital acquired infections. The objective of this study is to assess the neutrophil functional profiles and their associations with SSIs.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for an elective open gastrointestinal surgical procedure or spine fusion surgery

Exclusion Criteria:

* On chronic immunosuppressive drugs such as chronic corticosteroid use
* preexisting immunodeficiency diseases

Ages: 12 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients presenting for elective surgical procedures (open gastrointestinal surgery or spine fusion surgery) at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil populations | up to 3 days
  compare neutrophil population between patients with SSI and without SSI by delineating transcriptomic profiles
Neutrophil functional impairment | up to 3 days
  illustrate neutrophil subpopulation associated with neutrophil functional impairment and SSIs by probing phagocytosis and reactive oxygen species formation

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Yuki, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hopsital, Boston, Massachusetts, United States